CLINICAL TRIAL: NCT04249739
Title: Phase II Study of Pembrolizumab + Capecitabine／Oxaliplatin (CapeOx)(HER2 Negative ARM) or Pembrolizumab + Trastuzumab+ Capecitabine／Cisplatin (HER2 Positive ARM) in Metastatic GC as First-line Treatment
Brief Title: Pembrolizumab + Capecitabine／Oxaliplatin (CapeOx) -HER2 Nagative and Pembrolizumab + Trastuzumab + Cisplatin/Capecitabine HER2 Positive
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD, PhD,Principal Investigator, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-11-089
Record Dates: First submitted 2020-01-21; First posted 2020-01-31 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Assigned to 1 group according to the result of HER2. <Cohort A>: HER2 negative patients CapeOx+Pembrolizumab therapy (N=78)
  * Cycle 1 CapeOX
  * Cycle 2 up to Cycle 8 CapeOX + pembrolizumab therapy
  * Cycle 9 up to Cycle 35 Capecitabine + pembrolizumab therapy
    * CapeOx + Pembrolizumab administered until disease progression, unacceptable toxicity or patient's refusal.
      1. Cycle: Day 1 through Day 21)
  <Cohort B>: HER2 positive patients Cape/Cis+Trastuzumab+Pembrolizumab therapy (N=15)
  * Cycle 1 Capecitabine + cisplatin (Cape/Cis)
  * Cycle 2 up to Cycle 8 Cape/Cis + Trastuzumab + pembrolizumab therapy
  * Cycle 9 up to Cycle 35 Capecitabine + Trastuzumab + pembrolizumab therapy
    * Cape/Cis + Trastuzumab + Pembrolizumab administered until disease progression, unacceptable toxicity or patient's refusal.
      1. Cycle: Day 1 through Day 21)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CapeOx+Pembrolizumab(HER2 negative) (Experimental): <Cohort A>: HER2 negative patients CapeOx+Pembrolizumab therapy (N=78)
  * Cycle 1 CapeOX
  * Cycle 2 up to Cycle 8 CapeOX + pembrolizumab therapy
  * Cycle 9 up to Cycle 35 Capecitabine + pembrolizumab therapy
    * CapeOx + Pembrolizumab administered until disease progression, unacceptable toxicity or patient's refusal.
      1. Cycle: Day 1 through Day 21)
  Interventions: Drug: Pembrolizumab
- Cape/Cis+Trastuzumab+Pembrolizumab (HER2 positive ) (Experimental): Cape/Cis+Trastuzumab+Pembrolizumab therapy (N=15)
  * Cycle 1 Capecitabine + cisplatin (Cape/Cis)
  * Cycle 2 up to Cycle 8 Cape/Cis + Trastuzumab + pembrolizumab therapy
  * Cycle 9 up to Cycle 35 Capecitabine + Trastuzumab + pembrolizumab therapy
    * Cape/Cis + Trastuzumab + Pembrolizumab administered until disease progression, unacceptable toxicity or patient's refusal.
      1. Cycle: Day 1 through Day 21)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. Keytruda ™ (pembrolizumab) has recently been approved in the United Stated for the treatment of patients with unresectable or metastatic melanoma and disease progression following ipilimumab and, if BRAF V600 mutation positive, a BRAF inhibitor.
  Other Names: Keytruda; MK3475

SUMMARY:
This study is an open-label, single arm, phase II trial the efficacy and safety of pembrolizumab + CapeOx (HER2 negative ARM) or pembrolizumab + Trastuzumab + Capecitabine/Cisplatin (HER2 positive ARM) as first line therapy in advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma.

DETAILED DESCRIPTION:
Cohort A is allocated for the patients with Advanced Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma who confirmed with HER2 negative, and approximately 78 subjects will be enrollment to evaluate the efficacy and safety of pembrolizumab + Capecitabine/oxaliplatin.

Cohort B is allocated for the patients with Advanced Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma who confirmed with HER2 positive, and approximately 15 subjects will be enrollment to evaluate the efficacy and safety of pembrolizumab + Trastuzumab + Capecitabine/Cisplatin

(1 Cycle: Day 1 through Day 21)

Planned Biopsy Analysis immediate pre-treatment biopsy before chemotherapy; Newly-obtained specimens are defined as FFPE-preserved blocks or fresh tissue collected up to 12 weeks prior to C1D1.

2.on treatment primary tumor biopsy (C2D1 - 3 days window; before administration of C2D1) to explore whether tumor has change in characters (i.e., immune desert to immune infiltration) 3.on treatment primary tumor biopsy (C7D1 - 3 days window; before administration of C7D1) to explore whether tumor has change in characters (i.e., immune desert to immune infiltration) 4.At progression biopsy will be optional whenever the tumor biopsy is feasible.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial. The subject may also provide consent for Biomedical Research. However, the subject may participate in the main trial without participating in Biomedical Research.
2. Be 19 years of age on day of signing informed consent (or acceptable age according to local regulations, whichever is older).
3. Have histologically or cytologically-confirmed diagnosis of gastric or GEJ adenocarcinoma. (EBV positive GC and MSI-H GC will be excluded from this study). The patients must have EBV negative and MSS (or MMR-proficient) GC to enter this study.For cohort B, GC patients with HER2 + will be enrolled.
4. Be HER2-positive defined as either IHC 3+ or IHC 2+ in combination with ISH+ (or FISH), as assessed by central review on primary or metastatic tumor. ISH positivity is defined as a ratio of ≥ 2.0 for the number of HER2 gene copies to the number of signals for CEP17. If the ratio is <2.0 but the HER2 gene copy number is >6 the participant may be considered ISH-positive.
5. Have metastatic disease or locally advanced, unresectable disease.
6. Have measurable disease based on RECIST 1.1. as determined by investigator. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. Newly obtained fresh biopsy is required before enrollment (stomach biopsy required but if stomach cancer is not intact due to previous surgery, metastatic lesion biopsy can substitute)
8. Have a performance status of 0 or 1 on the ECOG Performance Scale.
9. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

111.Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication . Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

12.Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
3. squamous cell or undifferentiated gastric cancer.
4. Has pre-existing peripheral neuropathy >Grade 1.
5. Is a WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment . If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
6. Has active TB (Bacillus Tuberculosis)
7. Hypersensitivity to pembrolizumab or any of its excipients.
8. Has a known sensitivity to any component of oxaliplatin or xeloda
9. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
10. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
11. Has a known history of prior malignancy except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for 2 years since initiation of that therapy.
12. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
14. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis. Participants with asthma that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would not be excluded from the study.
15. Has an active infection requiring systemic therapy.
16. Has had an allogenic tissue/solid organ transplant.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
20. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
21. Has received prior therapy with an anti-HER2 agent.
22. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
23. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
24. Has received a live vaccine within 30 days of planned start of study therapy.
25. Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or staff directly involved with this trial, unless prospective IRB approval (by chair or designee) is given allowing exception to this criterion for a specific subject.
26. Participants with ascites if it needs draining within 2 weeks or diuretic within 2 weeks of consenting this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
ORR (objective response rate) per RECIST 1.1 | 24months
  Git is recommended that the subject bediscontinued from the study treatment unless, in the Investigator's opinion, the subject is deriving benefit from treatment.

SECONDARY OUTCOMES:
Genomic analysis | 24months
  Whole Exome Sequencing at baseline, RNA-seq pre and post

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lim SH, Kuwata T, An M, Hong JY, Kim ST, Matsubara Y, Shitara K, Lee J. Dynamic modulation of claudin18.2 expression and remodeling of the tumor microenvironment in gastric cancer during chemo-immunotherapy. J Immunother Cancer. 2025 Sep 29;13(9):e012683. doi: 10.1136/jitc-2025-012683. PMID 41027671